CLINICAL TRIAL: NCT04136717
Title: Influence of Automatic Oxygen Titration Device (FreeO2) on Percentage of Time Within Oxygen Saturation Target and Induced Hypercapnia During Noninvasive Ventilation for Patients Hospitalized for an Acute Exacerbation of COPD or a Bariatric Surgery
Brief Title: Influence of FreeO2 on Percentage of Time Within Oxygen Saturation Target Using Noninvasive Ventilation (NIV) and Continuous Positive Airway Pressure (CPAP) for Patients Admitted for AECOPD or Bariatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: François Lellouche (Other)
Responsible Party: Sponsor-Investigator, François Lellouche, Principal Investigator, Laval University
Organization: Laval University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2020-3275, 21796
Record Dates: First submitted 2019-10-15; First posted 2019-10-23 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: COPD Exacerbation; Oxygen Toxicity; Abdominal Obesity; Surgery
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COPD patients (Other): Patients with acute exacerbation of COPD and respiratory acidosis under oxygen therapy.
  Interventions: Other: Washout period; Device: NIV - FreeO2; Device: Nasal High flow Oxygen therapy - FreeO2
- Bariatric surgery patients (Other): Obese patients after gastric surgery under CPAP.
  Interventions: Other: CPAP - Oxygen constant flow; Other: CPAP - FreeO2

INTERVENTIONS:
Other: Washout period — During this period the patients will breath spontaneously oxygen titrated using the FreeO2 device with a SpO2 target set at 90%. The period duration is 30 minutes.
  Arms: COPD patients
Device: NIV - FreeO2 — During this period the patients will receive NIV using FreeO2 device for oxygen titration with a SpO2 target set at 90%. Initially, the inspiratory pressure will be set to obtain a tidal volume between 6 to 8 mL/Kg of predictive body weight and positive end-expiratory end pressure (PEEP) at 5 centimeters of water (cmH2O).
  After NIV initiation, the parameters can be adjusted to improve patient comfort. The period duration is 30 minutes.
  Arms: COPD patients
Device: Nasal High flow Oxygen therapy - FreeO2 — During this period the patients will receive NHFOT using the FreeO2 device for oxygen titration with a SpO2 target set at 90%. The high flow device will be set at 30 lpm.The period duration is 30 minutes.
  Arms: COPD patients
Other: CPAP - Oxygen constant flow — During this period, the patients will have their own CPAP with oxygen adjusted by hospital staff according to hospital protocol. The period duration is 15 minutes.
  Arms: Bariatric surgery patients
Other: CPAP - FreeO2 — During this period, the patients will have their own CPAP with oxygen adjusted using the FreeO2 device. SpO2 target will be set at 90% The period duration is 60 minutes.
  Arms: Bariatric surgery patients

SUMMARY:
The main objective is to evaluate the FreeO2 device combined with noninvasive respiratory support technique for COPD patients and postoperative bariatric surgery patients.

The main hypothesis is that FreeO2 device for oxygen therapy associated with NIV or nasal high flow oxygen therapy (NHFOT) allows to reach better oxygenation and avoid hypoxemia and hyperoxia.

DETAILED DESCRIPTION:
Bariatric surgery patients:

The main objective of this study is to evaluate the time spent in the SpO2 target (+/- 2% SpO2 target) and partial pressure of carbon dioxide (PCO2) values on patients with morbid obesity after bariatric surgery.

COPD patients:

The main objective of this study is to evaluate the time spent in the SpO2 target (+/- 2% SpO2 target) and PCO2 values on patients with exacerbation of COPD (hypercapnic patients) with different ventilatory supports (NIV and NHFOT) associated with FreeO2.

ELIGIBILITY:
Inclusion Criteria (AECOPD):

* Respiratory acidosis (pH <= 7.35 and PaCO2 > 45 mmHg), with or without NIV (last blood gas available during hospitalization)
* Oxygen therapy and/or SpO2 <90% room air (FiO2 <= 50% or nasal cannula <= 7 L/min to maintain SpO2 90%)
* High flow nasal cannula with flow <= 30 L/min

Inclusion Criteria (Bariatric surgery post-op):

* Patients using CPAP before the surgery (obstructive sleep apnea documented).
* Patients with obesity hypoventilation syndrome in addition to obstructive sleep apnea can be included.

Exclusion Criteria:

* Age < 18
* Pregnancy
* Respiratory distress or other clinical situation requiring continuous NIV or CPAP
* Glasgow < 12 or agitation/delirium/dementia (limiting NIV)
* Any contraindication to NIV (state requiring immediate endotracheal intubation, pneumothorax, recent esophagus surgery)
* Hemodynamic instability (at the beginning of the study) (increasing doses of vasopressors or inotropes)
* Refusal to consent to the study

  5 patient with AECOPD and 5 patient with bariatric surgery will be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of time within SpO2 target | AECOPD Patients: Day 1; Up to 120 minutes after start study procedures. Bariatric surgery patients: Day 1; up to 75 minutes after start study procedures(post-op).
  (SpO2 90 +/- 2%)

SECONDARY OUTCOMES:
Percentage of time in hypoxemia | AECOPD Patients: Day 1; Up to 120 minutes after start study procedures. Bariatric surgery patients: Day 1; up to 75 minutes after start study procedures(post-op).
  (SpO2 < -2% of SpO2 target)
Percentage of time in severe hypoxemia | AECOPD Patients: Day 1; Up to 120 minutes after start study procedures. Bariatric surgery patients: Day 1; up to 75 minutes after start study procedures(post-op).
  (SpO2 < -5% of SpO2 target)
Percentage of time in hyperoxia | AECOPD Patients: Day 1; Up to 120 minutes after start study procedures. Bariatric surgery patients: Day 1; up to 75 minutes after start study procedures(post-op).
  (> +5% of SpO2 target)
PCO2 value after each period | AECOPD Patients: Day 1; 30 minutes, 60 minutes, 90 minutes, 120 minutes after start study procedures. Bariatric surgery patient: Day 1; 15 minutes and 75 minutes after start study procedures.
  Measure PCO2 with blood gases after each period

CONTACTS AND LOCATIONS:
Locations (1):
- Institut universitaire de Cardiologie et de Pneumologie - Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No